CLINICAL TRIAL: NCT00624338
Title: A Randomised, Double-blind, Placebo Controlled, Multicentre Prospective Dose-finding Phase II/III Study With Atacicept Given Subcutaneously to Subjects Having Recently Experienced a Flare of Systemic Lupus Erythematosus (SLE)
Brief Title: Atacicept Phase 2/3 in Generalized Systemic Lupus Erythematosus (APRIL-SLE)
Acronym: APRIL-SLE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27646
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Atacicept 75 and 150 mg; Placebo
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Atacicept 75 mg (Experimental)
  Interventions: Drug: Atacicept 75 mg
- Atacicept 150 mg (Experimental)
  Interventions: Drug: Atacicept 150 mg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: Atacicept 75 mg — 75 milligram (mg) atacicept injection will be administered subcutaneously twice weekly during initial loading period for 4 weeks followed by once weekly during maintenance period for subsequent 48 weeks.
  Arms: Atacicept 75 mg
Drug: Atacicept 150 mg — 150 mg atacicept injection will be administered subcutaneously twice weekly during initial loading period for 4 weeks followed by once weekly during maintenance period for subsequent 48 weeks.
  Arms: Atacicept 150 mg
Other: Placebo Comparator — Placebo matched to atacicept injection will be administered subcutaneously twice weekly during initial loading period for 4 weeks followed by once weekly during maintenance period for subsequent 48 weeks.
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy and safety of atacicept compared to placebo in preventing new flares in subjects with systemic lupus erythematosus (SLE) and to confirm the optimal dose of atacicept for treatment of subjects with SLE and gain information on the effect of atacicept on markers specific to its mechanism of action (MoA) and their correlation to disease activity/progression. Study medication will be administered through subcutaneous (under the skin) injections, beginning with twice weekly injections for the first 4 weeks, followed by once weekly doses for 48 weeks. Following the last treatment, a safety follow-up period of 24 weeks will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 16 years of age or older
* Disease history of at least six months meeting at least 4 out of the 11 American College of Rheumatology (ACR) criteria for SLE
* Active SLE with at least one British Isles Lupus Assessment Group (BILAG) flare A or B at screening requiring a change in the dose of corticosteroids
* Positive antinuclear antibody (ANA) or anti-double-stranded deoxyribonucleic acid (dsDNA) at screening
* Female subjects must be willing to avoid pregnancy by using an adequate method of contraception for 4 weeks prior to Study Day 1, during the trial and 24 weeks after the last dose of study medication
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Active moderate to severe glomerulonephritis (kidney impairment) as defined in the protocol
* Active central nervous system SLE deemed to be severe/progressive and/or associated with significant cognitive impairment leading to inability to provide informed consent and/or comply with the protocol
* Previous treatment with rituximab, abatacept, or belimumab
* History of demyelinating disease such as multiple sclerosis (MS) or optic neuritis
* Other protocol defined exclusion criteria could apply

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2008-01; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (113):
- United States (18):
  - Division of Clinical Immunology and Rheumatology - UAB, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Research Site, San Diego, California
  - Inland Rheumatology Clinical Trials Inc, Upland, California
  - Research Site, Jacksonville, Florida
  - Research Site, Boise, Idaho
  - Brigham and Women's Hospital, Boston, Massachusetts
  - US Local Medical Information, Rockland, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Justus J. Fiechtner, MD, MPH, Lansing, Michigan
  - SUNY Health Science Center at Brooklyn, Brooklyn, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - Hospital for Special Surgey, New York, New York
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Division of Immunology, Cincinnati, Ohio
  - Research Site, Temple, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Quilmes
  - Research Site, San Juan
  - Research Site, San Miguel de Tucumán
- Australia (4):
  - Research Site, Cairns
  - Research Site, Clayton, Victoria
  - Research Site, Sunshine Coast, Queensland
  - Research Site, Woodville S.A.
- Research Site, Wein, Austria
- Research Site, Sofia, Bulgaria
- Croatia (4):
  - Research Site, Osijek
  - Research Site, Rijeka
  - Research Site, Split
  - Research Site, Zagreb
- Research Site, Prague, Czechia
- France (6):
  - Research Site, Bordeaux Pessac
  - Research Site, Lille
  - Research Site, Montpelier Cedex
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (7):
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Herne
  - Research Site, München
  - Research Site, Münster
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Research Site, Secunderabad, Andhra Pradesh, India
- Israel (4):
  - Research Site, Haifa
  - Research Site, Jerasalem
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
- Research Site, Riga, Latvia
- Research Site, Beirut, Lebanon
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Perak
  - Research Site, Seremban
- Mexico (2):
  - Research Site, Guadalajara Jalisco
  - Research Site, Tijuana, BC
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Leiden
  - Research Site, Maastricht
- Philippines (5):
  - Research Site, Angeles City, Pampanga
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Manila
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Szczecin
  - Research Site, Torun
  - Research Site, Warsaw
- Russia (7):
  - Research Site, Kemerovo
  - Research Site, Petrozavodsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tula
  - Research Site, Yaroslavl
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, New Belgrade
  - Research Site, Niška Banja
- South Africa (6):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Panorama, Western Cape
  - Research Site, Parlow, Western Cape
  - Research Site, Pinelands
  - Research Site, Stellenbosch, Western Cape
- South Korea (2):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santiago de Compostela
- Research Site, Sankt Gallen, Switzerland
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Ukraine (7):
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Ternopil
  - Research Site, Vinnytsia
  - Research Site, Zhytomyr
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Derived] Pitsiu M, Yalkinoglu O, Farrell C, Girard P, Vazquez-Mateo C, Papasouliotis O. Population pharmacokinetics of atacicept in systemic lupus erythematosus: An analysis of three clinical trials. CPT Pharmacometrics Syst Pharmacol. 2023 Aug;12(8):1157-1169. doi: 10.1002/psp4.12982. Epub 2023 Jun 18. PMID 37332136
- [Derived] Eslami M, Willen D, Papasouliotis O, Schuepbach-Mallpell S, Willen L, Donze O, Yalkinoglu O, Schneider P. Kinetics of free and ligand-bound atacicept in human serum. Front Immunol. 2022 Dec 2;13:1035556. doi: 10.3389/fimmu.2022.1035556. eCollection 2022. PMID 36532058
- [Derived] Isenberg D, Gordon C, Licu D, Copt S, Rossi CP, Wofsy D. Efficacy and safety of atacicept for prevention of flares in patients with moderate-to-severe systemic lupus erythematosus (SLE): 52-week data (APRIL-SLE randomised trial). Ann Rheum Dis. 2015 Nov;74(11):2006-15. doi: 10.1136/annrheumdis-2013-205067. Epub 2014 Jun 20. PMID 24951103

RESULTS

PARTICIPANT FLOW:
Groups:
- Atacicept 75 mg: 75 milligram (mg) atacicept injection was administered subcutaneously twice weekly during initial loading period for 4 weeks followed by once weekly during maintenance period for subsequent 48 weeks.
- Atacicept 150 mg: 150 mg atacicept injection was administered subcutaneously twice weekly during initial loading period for 4 weeks followed by once weekly during maintenance period for subsequent 48 weeks.
- Placebo: Placebo matched to atacicept injection was administered subcutaneously twice weekly during initial loading period for 4 weeks followed by once weekly during maintenance period for subsequent 48 weeks.
Period: Overall Study
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Started | 159 | 145 | 157
Treated | 157 | 144 | 154
Completed | 112 | 62 | 111
Not Completed | 47 | 83 | 46
Not completed — Adverse Event | 14 | 14 | 18
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 11 | 3 | 14
Not completed — Protocol Violation | 3 | 3 | 2
Not completed — Death | 0 | 2 | 0
Not completed — Immunoglobulin less than 3gram per liter | 1 | 0 | 0
Not completed — Termination of 150 mg group by Sponsor | 0 | 55 | 0
Not completed — Other | 15 | 5 | 9
Not completed — Randomized but not treated | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all the randomized participants, regardless of whether they received treatment.
Groups:
- Atacicept 75 mg: 75 mg atacicept injection was administered subcutaneously twice weekly during initial loading period for 4 weeks followed by once weekly during maintenance period for subsequent 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo | Total
Number analyzed (Participants) | 159 | 145 | 157 | 461
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (12.0) | 39.0 (12.8) | 39.0 (12.1) | 39.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 134 | 148 | 430
  Male | 11 | 11 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing a New Flare as Defined by British Isles Lupus Assessment Group (BILAG) Score A or B
Description: A flare was defined as having an adjudicated BILAG A or B score in any of the 8 organ systems during treatment, or imputed for participants who had premature treatment discontinuation. Discontinuations due to sponsor termination of the atacicept 150 mg group were not imputed as flares in this analysis. The BILAG disease activity index evaluates systemic lupus erythematosus (SLE) activity in 8 organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows. BILAG A: Disease sufficiently active requiring disease-modifying treatment (prednisone greater than 20 mg daily or immunosuppressants); BILAG B: Disease less active than in "A", mild reversible problems requiring only symptomatic therapy such as antimalarials, non-steroidal anti-inflammatory drugs (NSAIDs), or prednisone less than 20 mg day; BILAG C: Stable mild disease; BILAG D: System previously affected but now inactive; BILAG E: System never involved.
Time Frame: From screening up to Week 52
Population: Modified intent-to-treat (MITT) population included all the randomized participants who received study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 157 | 144 | 154
percentage of participants | 57.32 | 36.11 | 53.25
Statistical Analysis 1: Comparison: Atacicept 75 mg vs Placebo; Test type: Superiority or Other; p = 0.518, Regression, Logistic — Odds ratios were calculated from a logistic regression model adjusted for race and disease severity reported at screening; Odds Ratio (OR) = 1.160, 95% CI 2-sided [0.74 to 1.82]
Statistical Analysis 2: Comparison: Atacicept 150 mg vs Placebo; Test type: Superiority or Other; p = 0.003, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Atacicept 150 mg arm was discontinued prematurely. The analysis of 150 mg was considered post-hoc; Odds Ratio (OR) = 0.490, 95% CI 2-sided [0.31 to 0.78]

2. Secondary Outcome: Time to First New Flare as Defined by BILAG Score A or B
Description: A flare was defined as having an adjudicated BILAG A or B score in any of the 8 organ systems during treatment. Analysis was right-censored at Week 52. The hazard ratios and 95% confidence intervals were obtained from the Cox proportional hazards model. The 25th Percentile of time to new flare was reported using Kaplan-Meier estimates (Median was not reached). The BILAG disease activity index evaluates SLE activity in 8 organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows. BILAG A: Disease sufficiently active requiring disease-modifying treatment (prednisone greater than 20 mg daily or immunosuppressants); BILAG B: Disease less active than in "A", mild reversible problems requiring only symptomatic therapy such as antimalarials, NSAIDs, or prednisone less than 20 mg day; BILAG C: Stable mild disease; BILAG D: System previously affected but now inactive; BILAG E: System never involved.
Time Frame: From screening up to Week 52
Population: MITT population included all the randomized participants who received study treatment
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 157 | 144 | 154
days | 143 [112 to 226] | 310 [169 to NA] — Upper limit of confidence interval was not estimable as insufficient participants reached the event at the final time point for assessment. | 142 [87 to 197]
Statistical Analysis 1: Comparison: Atacicept 75 mg vs Placebo; Test type: Superiority or Other; p = 0.929, Regression, Cox — Cox proportional hazards model was performed to calculate hazard ratios and adjusted for race and disease severity at time of screening; Hazard Ratio (HR) = 0.984, 95% CI 2-sided [0.69 to 1.40]
Statistical Analysis 2: Comparison: Atacicept 150 mg vs Placebo; Test type: Superiority or Other; p = 0.009, Regression, Cox — [p-value comment as in outcome 2, analysis 1]; Atacicept 150 mg arm was discontinued prematurely. The analysis of 150 mg was considered post-hoc; Hazard Ratio (HR) = 0.562, 95% CI 2-sided [0.36 to 0.87]

3. Secondary Outcome: Percentage of Participants Experiencing a New Flare as Defined by BILAG Score A or B During Initial 24 Weeks
Description: A flare was defined as having an adjudicated BILAG A or B score in any of the 8 organ systems during treatment, or imputed for participants who had premature treatment discontinuation. The BILAG disease activity index evaluates SLE activity in 8 organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows. BILAG A: Disease sufficiently active requiring disease-modifying treatment (prednisone greater than 20 mg daily or immunosuppressants); BILAG B: Disease less active than in "A", mild reversible problems requiring only symptomatic therapy such as antimalarials, NSAIDs, or prednisone less than 20 mg day; BILAG C: Stable mild disease; BILAG D: System previously affected but now inactive; BILAG E: System never involved.
Time Frame: From screening up to Week 24
Population: MITT population included all the randomized participants who received study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 157 | 144 | 154
percentage of participants | 40.13 | 28.47 | 35.06
Statistical Analysis 1: Comparison: Atacicept 75 mg vs Placebo; Test type: Superiority or Other; p = 0.412, Regression, Logistic — Odds ratios were calculated from a logistic regression model, adjusted for race and disease severity reported at screening; Odds Ratio (OR) = 1.215, 95% CI 2-sided [0.76 to 1.94]
Statistical Analysis 2: Comparison: Atacicept 150 mg vs Placebo; Test type: Superiority or Other; p = 0.198, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Atacicept 150 mg arm was discontinued prematurely. The analysis of 150 mg was considered post-hoc; Odds Ratio (OR) = 0.722, 95% CI 2-sided [0.44 to 1.19]

4. Secondary Outcome: Percentage of Participants Within Ordinal Response Categories for British Isles Lupus Assessment Group (BILAG) Flares
Description: Ordinal response categories have been defined as: 1) No BILAG A, no BILAG B, and completed treatment, 2) No BILAG A, at least 1 BILAG B during treatment period, and 3) At least 1 BILAG A during treatment period. The BILAG disease activity index evaluates SLE activity in 8 organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows. BILAG A: Disease sufficiently active requiring disease-modifying treatment (prednisone greater than 20 mg daily or immunosuppressants); BILAG B: Disease less active than in "A", mild reversible problems requiring only symptomatic therapy such as antimalarials, NSAIDs, or prednisone less than 20 mg day; BILAG C: Stable mild disease; BILAG D: System previously affected but now inactive; BILAG E: System never involved.
Time Frame: Week 52
Population: MITT population included all the randomized participants who received study treatment. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 128 | 76 | 136
percentage of participants
  No BILAG A, no BILAG B, and completed treatment | 52.3 | 60.5 | 52.9
  No BILAG A, at least 1 BILAG B in treatment period | 39.8 | 28.9 | 38.2
  At least 1 BILAG A in treatment period | 7.8 | 10.5 | 8.8

5. Secondary Outcome: Mean Cumulative Corticosteroid Dose
Time Frame: Randomization up to Week 52
Population: MITT population included all the randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 157 | 144 | 154
mg | 2456.79 (1029.87) | 2018.87 (1062.61) | 2624.02 (812.44)

ADVERSE EVENTS:
Time Frame: Baseline up to 76 weeks (end of follow-up of the study)
Description: An adverse event (AE) is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 30/157 | 23/144 | 27/154
Other Adverse Events (participants affected / at risk) | 129/157 | 120/144 | 118/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atacicept 75 mg (N=157) | Atacicept 150 mg (N=144) | Placebo (N=154)
Pneumonia (Infections and infestations) | 5 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Bronchitis (Infections and infestations) | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 2
Abscess limb (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Leptospirosis (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Meningitis tuberculous (Infections and infestations) | 0 | 1 | 0
Mycetoma mycotic (Infections and infestations) | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Periproctitis (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Vasculitis gastrointestinal (Gastrointestinal disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chillblains (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Neuropsychiatric lupus (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 2
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Serum sickness (Immune system disorders) | 1 | 0 | 0
Biopsy cervix (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Social stay hospitalisation (Social circumstances) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atacicept 75 mg (N=157) | Atacicept 150 mg (N=144) | Placebo (N=154)
Upper respiratory tract infection (Infections and infestations) | 24 | 27 | 24
Urinary tract infection (Infections and infestations) | 22 | 23 | 17
Nasopharyngitis (Infections and infestations) | 21 | 16 | 11
Bronchitis (Infections and infestations) | 12 | 12 | 6
Sinusitis (Infections and infestations) | 8 | 4 | 10
Influenza (Infections and infestations) | 4 | 6 | 9
Injection site reaction (General disorders) | 16 | 22 | 3
Injection site erythema (General disorders) | 10 | 16 | 0
Pyrexia (General disorders) | 8 | 5 | 4
Injection site pruritus (General disorders) | 4 | 10 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 5 | 13
Nausea (Gastrointestinal disorders) | 11 | 7 | 6
Abdominal pain upper (Gastrointestinal disorders) | 8 | 3 | 3
Headache (Nervous system disorders) | 31 | 17 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 8
Hypertension (Vascular disorders) | 8 | 5 | 8
Hypotension (Vascular disorders) | 3 | 1 | 8

LIMITATIONS AND CAVEATS:
Atacicept 150 mg group was discontinued on 2 February 2011 based on the recommendation from the Independent Data Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other